CLINICAL TRIAL: NCT04641143
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Adjunctive Troriluzole in Obsessive Compulsive Disorder
Brief Title: Efficacy and Safety Study of Adjunctive Troriluzole in Obsessive Compulsive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV4157-302
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Troriluzole (Active Comparator): Troriluzole - 2 100mg capsules once daily for the first two weeks. Troriluzole - 2 140mg capsules once daily from week two through week ten.
  Interventions: Drug: Troriluzole
- Placebo (Placebo Comparator): Placebo - 2 100mg capsules once daily for the first two weeks. Placebo - 2 140mg capsules once daily from week two through week ten.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Troriluzole — Troriluzole - 2 100mg capsules QD for the first two weeks.
  Arms: Troriluzole
Drug: Placebo — Matching placebo - 2 140mg capsules QD from week two through week ten.
  Arms: Placebo

SUMMARY:
The study's purpose is to evaluate the efficacy and safety of troriluzole as adjunctive therapy compared to placebo in subjects with Obsessive Compulsive Disorder (OCD)

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of obsessive-compulsive disorder (OCD) as per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition as confirmed by the MINI at Screening; The duration of the subject's illness must be ≥ 1 year
2. An inadequate response to current Standard of Care medication defined as selective serotonin reuptake inhibitor (excluding fluvoxamine) or clomipramine treatment at an adequate and stable dose for at least 8 weeks prior to screening and at least 12 weeks at baseline (adequate dose defined by USPI labeling); an inadequate response as defined per the MGH-TRQ-OCD, there has been minimal or no meaningful clinical benefit as perceived by the subject
3. Determined by the investigator to be medically stable at baseline/randomization as assessed by medical history, physical examination, laboratory test results, and electrocardiogram testing. Subjects must be physically able and expected to complete the trial as designed

Exclusion Criteria:

1. Subjects with a history of more than two (2) previous failed or inadequate treatment classes given for an adequate duration at an adequate dose as defined by the MGH-TRQ-OCD.
2. Current or prior history of: bipolar I or II disorder, schizophrenia or other psychotic disorders, schizoaffective disorder, autism or autistic spectrum disorders, borderline personality disorder, antisocial personality disorder, Tourette's disorder, body dysmorphic disorder, hoarding disorder; or psychosurgery, Deep Brain Stimulation (DBS) or Electroconvulsive Therapy (ECT); or general medical condition that may confound safety and/or efficacy results
3. Previous treatment in a study with troriluzole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
The total score on the Yale-Brown Obsessive Compulsive Scale (YBOCS) | Change in total score from baseline, assessed at screening, baseline, week 4, 8 &10
  Improvement is measured by a lower total score

SECONDARY OUTCOMES:
Frequency of SAEs and AEs leading to discontinuation | From Screening through study completion, up to 10 weeks
  Percent difference between troriluzole vs placebo treatment emergent adverse events.
Improvement in functional disability as assessed by the change in Sheehan Disability Scale (SDS) | From baseline through study completion (up to 10 weeks)
  Change is measured as "mild" or "moderate" on the SDS
Improvement in global functioning responses assessed on the CGI-I scale. | From baseline through study completion (up to 10 weeks)
  Change is measured as "much improved" or "very much improved" on the CGII scale

CONTACTS AND LOCATIONS:
Locations (73):
- United States (73):
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - IMA Clinical Research, Phoenix, Arizona
  - NoeisisPharma, LLC, Phoenix, Arizona
  - CITrials (Clinical Innovations), Bellflower, California
  - Axiom Research, LLC, Colton, California
  - WR-PRI, LLC (Encino), Encino, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Clarity Clinical Research, Los Angeles, California
  - Excell Research, Inc, Oceanside, California
  - NRC Research Institute, Orange, California
  - Anderson Clinical Research, Redlands, California
  - Lumos Clinical Research Center, LLC, San Jose, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Stanford University, Stanford, California
  - Collaborative Neuroscience Research, Torrance, California
  - Yale University / Connecticut Mental Health Center, New Haven, Connecticut
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - Boca Raton Medical Institute, Boca Raton, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Research in Miami Inc, Hialeah, Florida
  - Accel Research Sites, Lakeland, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Health Care Family Rehab & Research, Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - FIRC, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - South Florida Research Phase I-IV , Inc., Miami Springs, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - APG Research, LLC, Orlando, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Omega Research Consultants, Orlando, Florida
  - MedBio Trials, Pembroke Pines, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Neurobehaviorial Institute, Weston, Florida
  - Conquest Research LLC, Winter Park, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - iResearch Savannah, Savannah, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Uptown Research Institute, Chicago, Illinois
  - Revive Research Institute, Elgin, Illinois
  - AMR-Baber Research, Inc, Naperville, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - CBH Health, Gaithersburg, Maryland
  - Pharmasite Research, Inc., Pikesville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Sisu at RMG, Springfield, Massachusetts
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Altea Research, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Integrative Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Bio Behavioral Institute, Great Neck, New York
  - Bioscience Research, LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Clinical Inquest Center, Ltd, Beavercreek, Ohio
  - Central States Research, LLC, Tulsa, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Comprehensive Psychiatric Care Providers, Providence, Rhode Island
  - BioBehavioral Research of Austin, Austin, Texas
  - Relaro Medical Trials, Dallas, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Mt.Olympus Medical Research LLC, Missouri City, Texas
  - Northwest Clinical Research Center, Bellevue, Washington